CLINICAL TRIAL: NCT04621370
Title: Priming the Tumour MicroEnvironment for Effective Treatment With Immunotherapy in Locally Advanced Rectal Cancer A Phase II Trial of Durvalumab (MEDI 4736) in Combination With Extended Neoadjuvant Regimens in Rectal Cancer
Brief Title: A Trial of Durvalumab (MEDI 4736) in Combination With Extended Neoadjuvant Regimens in Rectal Cancer
Acronym: PRIME-RT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liz-Anne Lewsley (Other)
Collaborators: University of Glasgow (Other); AstraZeneca (Industry); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor-Investigator, Liz-Anne Lewsley, Project Manager, Cancer Research UK, Glasgow
Organization: Cancer Research UK, Glasgow (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrimeRT-2018
Record Dates: First submitted 2020-10-19; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Rectal Cancer; Rectal Adenocarcinoma; Rectal Neoplasms
Keywords: Radiotherapy; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — durvalumab; Folfox protocol; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): * Durvalumab 1500mg IV over 60 minutes, starting in the week prior to day 1 of radiotherapy, and continuing every 4 weeks until completion of FOLFOX chemotherapy
  * Short course radiotherapy (25Gy delivered in 5 fractions) starting on day 1
  * FOLFOX chemotherapy will be given every 2 weeks, starting approximately 1-2 weeks after radiotherapy and continuing for 6 cycles in total
  * Assessment of response will be at approximately 16-18 weeks after day 1 of RT. If the patient is proceeding to surgery, this will be performed at approximately 18-20 weeks after day 1 of RT where possible.
  Interventions: Drug: Durvalumab; Drug: FOLFOX; Radiation: Short Course Radiotherapy (Arm A)
- Arm B (Active Comparator): * Durvalumab 1500mg IV over 60 minutes, starting in the week prior to day 1 of radiotherapy, and continuing every 4 weeks until completion of FOLFOX chemotherapy
  * Long course chemoradiotherapy (50Gy to boost volume, 45Gy to elective volume delivered in 25 fractions) starting on day 1
  * FOLFOX chemotherapy will be given every 2 weeks, starting approximately 1-2 weeks after radiotherapy for 4 cycles
  * Assessment of response at approximately 16-18 weeks after day 1 of RT. If the patient is proceeding to surgery, this will be performed at approximately 18-20 weeks after day 1 of RT where possible.
  Interventions: Drug: Durvalumab; Drug: FOLFOX; Radiation: Long course chemoradiation (Arm B); Drug: Capecitabine

INTERVENTIONS:
Drug: Durvalumab — Flat dose of 1500mg delivered intravenously over 30 minutes every 4 weeks.
  Other Names: MEDI 4736
Drug: FOLFOX — Oxaliplatin 85mg/m2 delivered intravenously as per institutional standard on Day 1 of mFOLFOX6 treatment every 2 weeks.
  5-fluorouracil bolus 400mg/m2 delivered intravenously as per institutional standard on D1 of mFOLFOX6 treatment every 2 weeks.
  5-fluorouracil infusion 2400mg/m2 delivered intravenously over 46 hours continuously as per institutional standard following bolus 5-fluorouracil.
  Other Names: mFOLFOX6
Radiation: Short Course Radiotherapy (Arm A) — 25 Gray of photon radiation treatment delivered over 5 fractions.
  Arms: Arm A
Radiation: Long course chemoradiation (Arm B) — 50 Gray of photon radiation treatment delivered over 25 fractions.
  Arms: Arm B
Drug: Capecitabine — Capecitabine is a non-cytotoxic pre-cursor of cytotoxic 5-fluorouracil and delivered in oral form. It is given concomitantly with long course radiation treatment on days of radiotherapy only. The dose is 825mg/m2 and this is delivered twice daily.
  Arms: Arm B

SUMMARY:
PRIME-RT is an open label, multi-centre phase II randomised trial with 1:1 allocation between arm A and arm B. The principal research question is whether the addition of durvalumab to FOLFOX chemotherapy and radiation treatment (either SCRT or LCRT) in the neoadjuvant setting for patients with locally advanced rectal cancer (LARC) improves rates of complete response. The working hypothesis is that the use of radiation and cytotoxic chemotherapy may prime the tumour immune microenvironment for treatment with immune checkpoint blockade. The main trial will commence after completion of a safety run-in which will enrol at least three patients per arm to test the safety and tolerability of the treatment combinations in each.

DETAILED DESCRIPTION:
In rectal cancer, strategies to enhance local treatment responses by expanding neoadjuvant regimens are sought to enable organ preservation in more patients. The addition of systemic FOLFOX post long course chemoradiotherapy (LCRT) and post short course radiotherapy (SCRT) has been reported with encouraging results demonstrating higher rates of complete response than with radiotherapy based treatment alone. Immunotherapy using PD-1/ PD-L1 inhibition is recognised to be effective in mismatch repair deficient colorectal cancer (dMMR). Generally, dMMR tumours are characterised by a higher mutational burden, a higher neoantigen load with high density T cell infiltrates and increased expression of PD-1/ PD-L1 in the tumour microenvironment (TME). Mismatch repair proficient (pMMR) colorectal cancer is not thought to be responsive to immunotherapies partly due to the fact they exhibit low levels of tumour infiltrating lymphocytes (TILs) and PD-1/PD-L1 within the TME. Attempts to expand the role of anti-PD-L1 treatment to pMMR CRC is likely to rely on provision of conventional DNA damaging treatments to increase tumour immunogenicity/ T cell infiltration. At baseline few rectal tumours (10-20%) demonstrate moderate-high grade CD3+ responses within the TME, but there is evidence that radiotherapy (e.g. SCRT or LCRT) and systemic chemotherapy (FOLFOX) induce favourable immune responses. In this phase II trial, the investigators plan to evaluate the potential treatment efficacy of anti-PD-L1 systemic anticancer treatment, durvalumab, alongside either SCRT or LCRT with FOLFOX in the gap up to post treatment assessment. This trial will evaluate rates of complete response in each arm as its primary endpoint in addition to safety and toxicity as secondary endpoints. It is a translationally rich trial which involves the collection of biospecimens prior to, during and following treatment in order to understand the molecular and immunological factors underpinning treatment response.

An initial 6 patient safety run-in (3 patients in each arm) will be performed treating patients with metastatic disease with a locally advanced rectal cancer in situ or patients with locally advanced rectal cancer who will never undergo radical surgery due to patient choice, in order to establish safety and lack of significant local toxicity due to the combination (for example colo-proctitis). Depending on the toxicity observed in the first 3 evaluable patients in each of the arm, an additional 3 patients may be add to that arm for the safety run-in cohort. Following an independent safety review and approval by an Independent Data Monitoring Committee (IDMC), the main trial will commence.

Following the safety run-in, 42 patients with non-metastatic, biopsy confirmed rectal adenocarcinoma (cT3b+, N+, EMVI+ based on MRI staging or low rectal tumours requiring abdominoperineal resection) will be recruited to the main trial and randomised to one of two treatment arms. These patients must have adequate physical fitness and no previous pelvic radiotherapy or immunotherapy.

Recruitment to the Safety Run-in period is expected to take 6 months (based on 6 patients in this cohort) with the main trial taking a further 12 months. Recruitment should therefore take place over a total period of 18 months. If the safety run-in requires more than 6 patients, these timelines will be revised. Patients will be followed up for 36 months from date of randomisation.

ELIGIBILITY:
Inclusion Criteria (Main trial):

1. Be willing and able to provide written informed consent for the trial.
2. Willingness to comply with scheduled visits, treatment plans and laboratory tests and other trial procedures including willingness to provide repeated biopsy samples of tumour via flexible sigmoidoscopy.
3. Age 18 or over on the day of signing informed consent.
4. Histologically confirmed non-metastatic, locally advanced rectal adenocarcinoma deemed appropriate for radical treatment.
5. Non-metastatic disease confirmed with CT of chest/abdomen and pelvis.
6. The rectal tumour must have at least one of the following high risk criteria on MRI scan:

   cT3b+ OR EMVI positive, OR Primary tumour or morphologically malignant lymph node at 2mm or less from the mesorectal fascia or beyond the mesorectal fascia OR Low rectal tumour and the consensus of the multi-disciplinary meeting is that abdomino-perineal excision would be required for sufficient surgical management.
7. ECOG performance status 0-1
8. No contra-indication to treatment with pelvic radiotherapy.
9. Primary disease which can be encompassed within a radical radiotherapy treatment volume.
10. Adequate haematological and biochemical function

Exclusion Criteria (Main trial):

1. Patients with Dihydroppyrimidine Dehydrogenase (DPD) deficiency (any degree).
2. Unable to have MRI assessment.
3. Patient weight less than or equal to 30kg.
4. Previous pelvic radiotherapy
5. Metastatic disease defined by CT (includes resectable metastases).
6. Previous treatment with immunotherapy.
7. Previous treatment with chemotherapy for the treatment of current malignancy or treatment with chemotherapy within the last 5 years for a separate malignancy (unless that malignancy was treated squamous/basal cell skin cancer, treated early stage cervical cancer or treated/biochemically stable, organ confined prostate cancer).
8. History of a separate malignancy in the last 5 years (other than treated squamous/basal cell skin cancer, treated early stage cervical cancer or treated/biochemically stable, organ confined prostate cancer).
9. Pregnant or lactating females or males unwilling to use a highly effective method of contraception. Women of childbearing potential, and men with female partners of childbearing potential, must agree to use adequate contraceptive measures (see section 9.1.12) for the duration of the study and for 6 months after the completion of study treatment.
10. Major surgery within 28 days prior to trial entry
11. Prolongation of corrected QT (QTc) interval to >470 msec when electrolyte balance is normal.
12. If a patient has had a recent occurrence (within 3-6 months) of a major thromboembolic event, such as pulmonary embolism or proximal deep vein thrombosis, they must be stable on therapeutic anticoagulation. Subjects with a history of clinically non-significant thromboembolic events, not requiring anticoagulation, are allowed on study.
13. Active inflammatory bowel disease affecting the colon and rectum based on previous endoscopy and defined as active by ongoing drug treatment.
14. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., levothyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
15. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisolone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial drug.
16. Has a history of (non-infectious) interstitial pneumonia or pneumonitis that required steroids or current pneumonitis.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Has received a live vaccine within 30 days prior to the first dose of trial drug. 21. Any patients receiving treatment with brivudine, sorivudine and analogues or patients who have not stopped these drugs at least 4 weeks prior to start of study treatment 22. Any patient with severe diarrhoea (defined as ≥ grade 3 diarrhoea despite maximum supportive measures and exclusion of underlying infection).
20. Known hypersensitivity for any component of any study drug.
21. Administration of any investigational drug within 28 days or 5 half-lives, whichever is longer, prior to receiving the first dose of trial treatment.
22. Uncontrolled Chronic Heart Failure (CHF), or history of myocardial infarction (MI), unstable angina, stroke, or transient ischemia within previous 6 months.
23. Patients with known malabsorption or inability to comply with oral medication.
24. Patients with known human immunodeficiency virus (HIV1/2). This is an exclusion criteria because the blood samples from these patients cannot be processed at the translational laboratories linked with this trial. Screening for HIV is not required for this trial.
25. Patients with known Hepatitis B or Hepatitis C. This is an exclusion criteria as the blood samples from these patients cannot be processed at the translational laboratories linked with this trial. Screening for hepatitis B or C is not required for this trial.
26. Receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment. Includes prior organ transplantation including allogenic stem-cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-12-07 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response | 6 months
  Pathological or clinical complete response

SECONDARY OUTCOMES:
Adverse events | During neo-adjuvant treatment and for up to at least 90 days after the last dose of Investigatinal Medicinal Product (IMP).
  Occurrence of Grade 3-5 treatment-emergent adverse events and treatment-related adverse events.
CD3+ T cell infiltrate | Week 2, week 6 and end of treatment (Week 15-18)
  Presence of a moderate-high grade CD3+ T cell infiltrate on rectal tumour biopsy during treatment.
Neoadjuvant Rectal (NAR) score | Immediately after the surgery
  In patients who do not achieve a clinical complete respose (cCR), the proportion of patients with a Neodjuvant Rectal (NAR) score <8. The NAR score is a pseudo-continuous scale with 24 possible discrete scores ranging from 0-100. A low score was defined as <8, intermediate as 8-16 and high as >16 with corresponding 5 year OS in this patient cohort of 92%, 89% and 68% respectively, showing that higher scores are associated with poorer prognosis.
MRI defined tumour regression | End of Treatment (Week 15-18)
  Proportion of patients achieving MRI-confirmed near or complete tumour regression
MRI defined down-staging | End of Treatment (Week 15-18)
  Proportion of patients achieving MRI-confirmed down-staging in T stage
Tumour regrowth | Through study completion, up to 36 months post randomisation
  Proportion of patients with local regrowth after a cCR.
Survival | 36 months
  Overall survival
Recurrence | 36 months
  Recurrence free survival
Colostomy | Immediately after surgery / throughout study completion, up to 36 months post randomisation
  Proportion of patients who have a permanent colostomy.
Delivery of radical treatment | End of treatment (Week 15-18)
  Proportion of patients who proceed to surgery (or who have a complete clinical response and go onto the deferred surgery pathway).
Radiotherapy delivery | End of treatment (Week 15-18)
  Proportion of patients receiving at least 4 fractions of short course RT or 20 fractions of long course RT.
Surgical complications | Immediately after surgery
  Proportion of patients with Grade 3-5 complications
European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 (EORTC QLQ-C30) | Baseline and months 3, 6, 12, 18, 24 and 30.
  EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, and social) (higher score = better functioning), global health status (higher score=better functioning), symptom scales (fatigue, pain, nausea/vomiting) (higher score= worse symptoms), and other (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties) (higher scores=worse difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer 29 (EORTC QLQ-CR29) | Baseline and months 3, 6, 12, 18, 24 and 30.
  All scales and single-item measurements range from 0 to 100. A higher score for a symptom scale / item indicates a higher symptomatology and problem level.
Euro Qol-5 dimensions 3 levels (EQ5D-3L) | Baseline and months 3, 6, 12, 18, 24 and 30.
  Quality of life questionnaire that measures quality of life in 5 dimensions on a 3 part scale (1=no problems, 3=extreme problems). Min score: 11111 Max score: 33333

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanna CR, O'Cathail SM, Graham JS, Saunders M, Samuel L, Harrison M, Devlin L, Edwards J, Gaya DR, Kelly CA, Lewsley LA, Maka N, Morrison P, Dinnett L, Dillon S, Gourlay J, Platt JJ, Thomson F, Adams RA, Roxburgh CSD. Durvalumab (MEDI 4736) in combination with extended neoadjuvant regimens in rectal cancer: a study protocol of a randomised phase II trial (PRIME-RT). Radiat Oncol. 2021 Aug 26;16(1):163. doi: 10.1186/s13014-021-01888-1. PMID 34446053